CLINICAL TRIAL: NCT06494163
Title: Exercise Training in Women With Heart Disease: A Randomized Controlled Trial
Brief Title: Exercise Training in Women With Heart Disease 2
Acronym: EXCEED2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20240363-01H
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases; Coronary Heart Disease
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care + moderate-intensity continuous exercise training (Experimental): 2 days/week Warm-up: 60-70% peak HR - 10min Training: 70-85% peak HR - 35min Cool-down: 60-70% peak HR - 15min
  Interventions: Behavioral: Exercise
- standard care + high-intensity interval training (Experimental): 2 days/week Warm-up: 60-70% peak HR - 10min Training: 85-95% peak HR - 25 minutes (4x4-minutes of high-intensity intervals interspersed with 3 minutes of low-intensity intervals) Cool-down: 60-70% peak HR - 10min
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — The MICT and HIIT intervention groups will complete supervised virtual exercise sessions for 12 weeks using Zoom care or Microsoft Teams as a backup resource. The appointments will be scheduled and conducted 2 days per week. Initially, exercise intensity will be determined from participants' peak HR achieved during a baseline CPET.

SUMMARY:
This study will compare the effects of two different types of training on exercise capacity in women with coronary heart disease (CHD). Participants will be randomized into either the virtual high-intensity interval training (HIIT) or the virtual moderate-to-vigorous intensity continuous training (MICT). After randomization, patients will exercise twice a week, for 12 weeks. The sessions will be conducted virtually. Patients will undergo a maximal exercise test, cardiometabolic indicators (height (cm), body mass (kg), body composition (%), waist circumference (cm) and, resting blood pressure) and complete questionnaires about quality of life, mental health, self-determined motivation, self-efficacy and enjoyment.

DETAILED DESCRIPTION:
Heart disease is a leading cause of death for women. Women who suffer a heart attack are more likely than men to be inactive, have lower fitness, and die in the next year; patients also report poor mental health and quality of life (QoL), and have a greater risk of cardiovascular disease risk factors. This clinical research project is concerned about women with heart disease and how to improve their fitness, mental health, and QoL using a different kind of exercise. Currently, moderate-to-vigorous intensity continuous training, MICT, is the most frequently prescribed for women with heart disease. Unfortunately, this exercise tends to be a burden and is time-consuming. The study aims to test if high-intensity interval training (HIIT, alternating periods of hard exercise and rest) is better than MICT at improving fitness, mental health, QoL, and exercise dedication in women with heart disease. The investigators will recruit 104 women with heart disease. The investigators will first assess the health measures outlined above and then randomly assign people to MICT or HIIT. Both groups will attend virtual exercise sessions 2 days/week for 12 weeks. The MICT group will perform Zumba/movement-based exercise for 35 minutes at an intensity level of 70-85% of their maximal effort. The HIIT group will perform Zumba/movement-based exercise for 25-minutes: this will consist of 4 periods of exercising for 4-minutes at an intensity level of 85-95% of their maximal effort, separated by 3 minutes of rest between each period. The investigators will assess the health measures again after 12 and 26 weeks. The scores for people in the two groups will then be compared. HIIT has never been evaluated as an alternative for MICT in a large women-only group with heart disease. If this clinical trial shows that HIIT helps these women improve their physical and psychosocial health over usual practice, then health care professionals caring for women with heart disease will have an alternative, effective treatment option to provide women in need.

ELIGIBILITY:
Inclusion Criteria:

1. Women (i.e., female sex assigned at birth) with CHD (e.g., coronary artery bypass grafting surgery [CABG], percutaneous coronary intervention [PCI], acute myocardial infarction [MI], MI with no obstructive coronary artery disease [MINOCA], or ischemia with no obstructive coronary artery disease [INOCA] at least 4 weeks post procedure or event; based on clinical evidence this is a safe period of time to exercise);
2. Patient is able to perform a symptom limited CPET (this is the primary outcome and needed to determine peak HR for the exercise training prescription); and
3. Patient is able to read and understand English or French.

Exclusion Criteria:

1. Patient is currently participating in routine exercise training (>2x/week, routine exercise training is defined as a planned, structured, and repetitive exercise that is performed in order to maintain or improve physical fitness.) (this may reduce the impact of HIIT or MICT on outcomes);
2. Patient has: NYHA class III-IV heart failure symptoms; unstable angina; or established diagnosis of chronic obstructive pulmonary disease, severe mitral or aortic stenosis, or hypertrophic obstructive cardiomyopathy (this may interfere with the ability to engage in MICT or HIIT);
3. Patient has uncontrolled arrhythmia (this may impact the HR-based exercise training prescription and monitoring);
4. Patient is unable to provide written informed consent; or
5. Patient is unwilling or unable to return for follow-up visits at 12 and 26 weeks.
6. Patient is unwilling to be randomized to HIIT or MICT.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants whose gender identity may differ from their birth-assigned sex (female) will be considered eligible for the study
Enrollment: 172 (Estimated)
Dates: Start 2024-08-12 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | from baseline to week-6 and from baseline to week-12
  will be measured using a gold standard symptom-limited, cardiopulmonary exercise test (CPET) on a treadmill (or on an alternate equipment, such as a cycle ergometer or recumbent bike). Gas exchange will be monitored continuously (- Parvo Medics TrueOne® 2400); the highest 20 second average rate of oxygen uptake achieved (i.e. peak VO2 in mL/kg/min) during the last minute of the CPET will represent exercise capacity.

SECONDARY OUTCOMES:
physical and mental health | from baseline to 12 weeks and baseline to 26 weeks
  hysical and mental health will be measured using the Mental Health Composite Scale (MCS) and Physical Composite Scale (PCS) of the Short Form-36 questionnaire. It consists of 36 items that contribute to eight subscales summarized into a physical component summary scale (PCS) and a mental component summary scale (MCS). A higher score on a 0-100 scale indicates a better quality of life.
Disease-specific Quality of Life, global health, physical and emotional health | from baseline to 12 weeks and baseline to 26 weeks
  measured using the HeartQoL, a validated 14-item questionnaire that assesses patients' feelings on how heart disease affects daily functioning, providing a global-health related QoL score and physical and emotional subscales. Higher score means better quality of life. Score range from 0-3, where higher scores represents better heart quality of life.
Anxiety symptoms | from baseline to 12 weeks and baseline to 26 weeks
  assessed with the Generalized Anxiety Disorder-7 (GAD-7).Participants rate statements regarding symptoms of anxiety on a 4-point scale (0=not at all; 4=nearly every day). The items are summed to obtain a score ranging from 0-21.
Depressive symptoms | from baseline to 12 weeks and baseline to 26 weeks
  Depressive symptoms: assessed with the Patient Health Questionnaire (PHQ-9), a 9-item scale based on diagnostic criteria for depressive disorders. Participants rate statements on a 4-point scale (0=not at all; 4=nearly every day), yielding a single score indicating severity of depression symptoms.
body composition - BMI | from baseline to 12 weeks and baseline to 26 weeks
  body mass (kg) and height (cm) will be measured to calculate body mass index (kg/m^2)
body composition - Waist circumference | from baseline to 12 weeks and baseline to 26 weeks
  Changes in body composition from baseline to 12 weeks and baseline to 26 weeks are measured by waist circumference (cm).
body composition - BIA | from baseline to 12 weeks and baseline to 26 weeks
  Changes in body composition from baseline to 12 weeks and baseline to 26 weeks are measured by bioelectrical impedance (%)
Vital Signs - Resting Blood Pressure | from baseline to 12 weeks and baseline to 26 weeks
  changes in vital signs will be measured using resting blood pressure (mmHg) in a seated position after a 5-minute rest period on the right arm using an automated monitor (BPTru) that measures 3 times at 2-minute intervals.
Vital Signs - Resting Heart Rate | from baseline to 12 weeks and baseline to 26 weeks
  changes in vital signs will be measured using resting heart rate (bpm)
Self-determined motivation for exercise | from baseline to 12 weeks and baseline to 26 weeks
  the 24-item Behavioural Regulation in Exercise questionnaire (BREQ-3) yields an overall Relative Autonomy Index (RAI) score, representing overall self-determined motivation. The scale ranges from -3 "amotivation to +3 "intrinsic regulation".
Overall self-efficacy for exercise | from baseline to 12 weeks and baseline to 26 weeks
  the 9-item Multidimensional Self-Efficacy for Exercise Scale (MSES-R) yields an overall self-efficacy for exercise score reflecting scheduling, task and coping self-efficacy. The MSES consists of nine items on a 100% confidence scale ranging from 0 = "no confidence" to 100 = "completely confident."
physical activity enjoyment | from baseline to 12 weeks and baseline to 26 weeks
  the 18-item Physical Activity Enjoyment Scale (PACES) measures the extent (on a 7-point Likert scale) to which participants enjoy doing physical activity. Overall enjoyment for physical activity score is determined by summing the items, with a range of 18-126 being possible. Higher scores indicate higher enjoyment.
Gender | from baseline to 12 weeks and baseline to 26 weeks
  assessed using the Genesis-Praxy questionnaire.

OTHER OUTCOMES:
Physical activity levels | from baseline to 12 weeks and baseline to 26 weeks
  will be measured objectively. The ActiGraph wGT3X-BT accelerometer (ActiGraph, Pensacola, Florida) will be worn over the right hip for 7 days
Program compliance | from baseline to 12 weeks
  Staff will record the number of MICT or HIIT sessions attended over the 12-week period (attended/prescribed x 100 = % compliance). Staff will record the number of MICT or HIIT sessions attended over the 14 weeks of unsupervised virtual exercise session.
  Reasons for missing exercise sessions and program drop-out will be collected to inform the development of strategies to engage women in CR.
Participant Experience | at 12 weeks
  As per the ORBIT model166 for developing effective behavioural treatments for chronic diseases, semi-structured focus groups (N=4)167 with patients (N=20, purposively selected according to age, gender, and medical conditions)168 will be conducted at 12 weeks to explore factors influencing adherence and satisfaction with MICT or HIIT. Each focus group will be 60-90 minutes in duration and will be held at times convenient for the participants
Feeling Scale | during intervention
  To assess affective response during exercise, the Feeling Scale will be completed during and immediately post exercise. The patient will report the value in a one-on-one chat function. The FS is an 11-point, single-item, bipolar rating scale commonly used for the assessment of affective valence (i.e., please-displeasure) during exercise. The scale ranges from -5 ("Very Bad") to +5 ("Very Good").
Participant Feedback | from baseline to 12 weeks
  To assess the participant's experience using a virtual intervention method.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reed, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided